CLINICAL TRIAL: NCT02069990
Title: Controlled, Randomized, Four-arm Comparative, Open Label, Multi-centric Clinical Trial to Compare the Efficacy and Safety Parameters of the Once-a-week or Once-a-month Administered 7000 IU, or 30000 IU Vitamin D (Cholecalciferol) to a 1000 IU Dosage Applied Daily in Vitamin D Deficient Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Semmelweis University (Other)
Collaborators: Pharma Patent Kft. (Unknown)
Responsible Party: Principal Investigator, Istvan Takacs, university docent, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PAT12-730DS
Record Dates: First submitted 2014-02-18; First posted 2014-02-24 (Estimated); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 30000 IU cholecalcipherol once a week (Active Comparator): 30000 IU cholecalcipherol once a week oral
  Interventions: Drug: Cholecalciferol
- 7000 IU cholecalcipherol once a week (Experimental): 7000 IU cholecalcipherol once a week oral
  Interventions: Drug: Cholecalciferol
- 30000IU cholecalcipherol once a month (Experimental): 30000IU cholecalcipherol once a month oral
  Interventions: Drug: Cholecalciferol
- 1000 IU cholecalciferol once a day (Active Comparator): 1000 IU cholecalciferol once a day
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol

SUMMARY:
Circa-annual variations in 25-hydroxyvitamin D [25(OH)D] levels have been well established, and there also seems to be an effect of season on bone turnover and bone mass. been shown that bone turnover follows a circa-annual rhythm. On the basis of human clinical results, it was suggested that adipose tissue functions as a vitamin D buffering system that to a certain extent prevents uncontrolled synthesis of 25(OH)D in the liver. Directly related to this issue is the question of how much vitamin D is needed to ensure target serum 25-hydroxyvitamin D [25(OH)D] concentrations. According to the recommended dietary allowances, persons should achieve "levels of intake of essential nutrients considered to be adequate to meet the known nutritional needs of practically all healthy persons" Moreover it is important to note that the significant percentage of the population is temporarily of continuously deficient in vitamin D. In the similar condition of vitamin D deficiency, the aetiology is very different since only as almost exclusively as a consequence of a primary disease in children it is manifested: hypovitaminosis D is highly prevalent among children on renal substitution therapy, regardless of the type of therapy used and the stage of renal failure.

The rationale providing high dose strengths of vitamin D based on an assumption of better compliance especially in adult with senior age patients; also a potential for faster resolution of vitamin D deficiency, since utilization of cholecalciferol is higher when patients had low levels of 25(OH)D, and vice versa, there is a plateau phase when close to normal range (Vieth 2001).

According to clinical data, a doses equivalent of daily 1000 IU, (7000 IU per week, or 30000 IU per month) is considered as a minimal effective dose to treat vitamin D deficiency. The treatment of vitamin D with a duration of 30 days may result and increase of 6-12.5 nmol/L. With the deficiency criteria considered as <20 ng/ml, the vitamin supplementation is indicative, the treatment dosages should be adjusted to the increase planned to achieve the mid-normal range.

As the base of calculations, the doses of 40 IU results in an increase of 0.4 ng/ml in a period of 60 days. Accordingly 1000 IU in a period of 2-5 month resulted in an increase of approx 10 ng/ml. The risk of overdose in relatively low, since the absorption and the metabolic path is well controlled: automatic mechanisms downregulation at normal ranges.

In this study the there are three groups in the similar daily dose equivalent of 1000 IU/day. The absorption of daily , weekly and monthly dosing should have a buffered effect due to the body adipose tissues, balancing the daily 1,25(OH)D levels, and moreover to provide a biological reservoir. The three doses are considered as comparable in efficacy and safety.

The fourth group is intended to utilize the expanded dose range of 4286 IU/ day, using the 30.000 IU tablets on a weekly dosing schedule. This group is to demonstrate the efficacy of higher doses to normalize the vitamin D levels, within a reasonable timeframe of 60-90 days.

ELIGIBILITY:
Inclusion Criteria:

Subject are included as 18 years or older ( adults) with the following specific criteria:

* 25(OH)D level < 50 nmol/L (20 ng/ml)
* female subjects either postmenopausal status or under proper (continuous) contraception during the course of the study are allowed to be enrolled
* Subject informed willing to participate and ICF signed and dated properly

Exclusion Criteria:

* hypercalcaemia/ se Ca levels out of 2.20-2.60 mmol/L range
* symptoms or lab results of elevated se Ca during the last year
* hypercalciuria within the last two years
* renal stones formation in anamnesis
* sever kidney disease ( CKD 3 or higher grade)
* chronic or serious illness that may result in malabsorption, the metabolisms of vitamin D or bones
* severe grade of metabolic diseases, bone disorders, excluded the primary age related osteoporosis,
* obesity ( BMI>35)
* diseases that resulted in changed absorption of calcium
* CHF or angina pectoris,
* recent (<3 month) surgical traumatic treatment
* alcohol or drug abuse,
* Vitamin D therapy or food supplements applied with the last 2 months, (at 1000 IU or above)
* planned travel (more than 5 days-long to a region of high natural UVB exposition)
* regular ( >2 per month) artificial UVB exposition (solarium)
* permanent use of non-permitted concomitant medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2013-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Serum 25-OH-Vitamin-D level | 12 weeks
  Based on the changes in 25(OH)D versus to baseline, in each group, and compared to the group of 1000 IU daily dosage applied.
  1000 IU /day vs. 7000 IU/ week, eqv. 1000 IU/ day vs 30000 IU/ month egv. 1000 IU /day vs 30000 IU/week: superiority

SECONDARY OUTCOMES:
number of adverse events | 12 weeks
  Frequency of adverse events for each group compared to group "A" ( as standard 1000 IU/day therapy). Evaluation of adverse event includes patient reported symptoms and safety laboratory (seCa, seP, se creatinine, urinary Ca) abnormalities.
Serum PTH | 12 weeks
Urinary calcium | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lakatos, professor, Principal Investigator — Semmelweis University
Locations (2):
- Hungary (2):
  - Semmelweis University 1st Dept. of Int. Med-, Budapest
  - Ambulatory Dept of Józsefváros Health Services, Budapest

REFERENCES:
- See also: Related Info — http://www.akademiai.com/content/e5x1v473712727t3/